CLINICAL TRIAL: NCT00908388
Title: Evaluation of the GORE Conformable TAG® Thoracic Endoprosthesis for Treatment of Acute Complicated Type B Aortic Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAG 08-01
Record Dates: First submitted 2009-04-03; First posted 2009-05-25 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Type B Aortic Dissection
Keywords: Acute, Complicated Type B Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GORE Conformable TAG® Device Surgical Implant (Experimental)
  Interventions: Device: GORE TAG® Thoracic Endoprosthesis

INTERVENTIONS:
Device: GORE TAG® Thoracic Endoprosthesis — Endoprosthetic Implant

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of the GORE Conformable TAG Thoracic Endoprosthesis (CTAG) for treatment of subjects with acute complicated type B aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of acute complicated type B aortic dissection:

   * Dissection is acute Time from symptom onset to dissection diagnosis ≤14 days
   * Dissection is complicated

   Subject must present with at least one of the following:
   * Rupture in the setting of an aortic dissection defined as hemorrhage outside of the aortic boundaries -which is noted by CT scan (hemorrhage must be differentiated from reactive effusions by the investigator, or if equivocal, having elevated Hounsefield units as determined by the radiologist).
   * Clinical evidence of malperfusion, in the setting of an aortic dissection, defined as:

     * Clinical or radiographic evidence of visceral hypoperfusion.
     * Clinical or radiographic evidence of renal hypoperfusion.
     * Clinical or radiographic evidence of lower extremity hypoperfusion.
     * Clinical or radiographic evidence of spinal cord hypoperfusion.

       * Dissection is type B Entire dissection is distal to the left subclavian artery
       * Primary Treatment Indication is Class 1 Aortic Dissection 46 Classical aortic dissection with intimal flap between true and false lumen with double barrel flow in thoracic aorta
       * Subjects with multiple entry tears are allowed to be enrolled in the study
2. Age 18 to 80 years
3. Primary treatment is endovascular treatment with the CTAG device. Adjunctive treatments may include left subclavian artery revascularization, percutaneous fenestration, aortic stenting, peripheral vessel stenting, surgical fenestration, and/or peripheral artery bypass
4. Proximal landing zone characteristics include:

   * Proximal extent of intended proximal landing zone cannot be dissected
   * Length ≥ 2.0 cm proximal to the primary entry tear
   * Trans-aortic diameter at proximal extent of intended landing zone between 16-42 mm (diameter assessed by flow lumen and thrombus, if present; calcium excluded)
   * Cannot be aneurysmal, heavily calcified, or have excessive intraluminal thrombus
   * Must be native aorta
   * May include left subclavian artery, if necessary
5. Subject is capable of complying with protocol requirements, including follow-up
6. Informed Consent Form is signed by subject or legal representative

Exclusion Criteria:

1. Primary treatment indication is Class 2-5 aortic dissection (intramural hematoma, limited dissection, penetrating atherosclerotic ulcer, iatrogenic dissection, traumatic dissection) 46
2. Concomitant aneurysm/disease of the ascending aorta, aortic arch, or abdominal aorta requiring repair (dissection extension into the abdominal aorta is acceptable)
3. Prior repair of DTA
4. Infected aorta
5. Subject has a systemic infection and may be at increased risk of endovascular graft infection
6. Persistent refractory shock (systolic blood pressure <90 mm Hg)
7. Bowel necrosis (Bowel necrosis will be characterized by direct observation with surgical exploration, or elevated serum lactate level and CT findings of portal venous gas, free intra-abdominal gas, pneumatosis intramural gas, and poor mucosal enhancement of thickened bowel wall)
8. Renal failure , defined as baseline creatinine ≥ 2.5 mg/dl
9. ASA risk classification = V (Moribund patient not expected to live 24 hours with or without operation)
10. Pregnant female
11. Major surgery within 30 days of treatment (other than left subclavian artery bypass or transposition)
12. Degenerative connective tissue disease, e.g., Marfan or Ehler-Danlos Syndrome
13. Treatment in another drug or medical device study within 1 year of study enrollment
14. History of stimulant abuse, e.g., cocaine or amphetamine, within 1 year of treatment
15. Tortuous or stenotic iliac and/or femoral arteries and the inability to use a conduit for vascular access
16. Planned coverage of left carotid or celiac arteries with the CTAG device
17. The planned endovascular procedure involves alterations to the CTAG device
18. Subject has known sensitivities or allergies to the device materials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cambria, MD, Principal Investigator — Massachusetts General Hospital
Locations (34):
- United States (34):
  - Birmingham, Alabama
  - Los Angeles, California
  - San Francisco, California
  - Stanford, California
  - Torrance, California
  - Gainesville, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Plymouth, Minnesota
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Albany, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - Houston, Texas
  - Temple, Texas
  - Charlottesville, Virginia
  - Madison, Wisconsin

REFERENCES:
- [Derived] Panthofer AM, Olson SL, Harris DG, Matsumura JS. Derivation and validation of thoracic sarcopenia assessment in patients undergoing thoracic endovascular aortic repair. J Vasc Surg. 2019 May;69(5):1379-1386. doi: 10.1016/j.jvs.2018.08.180. Epub 2018 Dec 28. PMID 30598352

RESULTS

PARTICIPANT FLOW:
Groups:
- GORE Conformable TAG® Device Surgical Implant: Subjects with acute complicated type B aortic dissection prospectively treated with endovascular surgery to implant the GORE ConformableTAG® Thoracic Endoprosthesis via femoral access. (permanent implant)
Period: Overall Study
Arm/Group | GORE Conformable TAG® Device Surgical Implant
Started | 50
Completed | 40
Not Completed | 10

BASELINE CHARACTERISTICS:
Groups:
- GORE Conformable TAG® Device Surgical Implant: Subjects prospectively treated with the GORE Conformable TAG® Thoracic Endoprosthesis for acute complicated type B aortic dissection
Arm/Group | GORE Conformable TAG® Device Surgical Implant
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality Incidence Through 30 Days Post-treatment
Time Frame: 30 Days Post-Treatment
Population: All subjects were analyzed. One subject whose vital status could not be confirmed was included as a death in this analysis.
Measure: Number; unit: participants
Arm/Group | GORE Conformable TAG® Device Surgical Implant
Number analyzed (Participants) | 50
participants | 5
Statistical Analysis 1: Comparison: GORE Conformable TAG® Device Surgical Implant; Test type: Superiority or Other; p = .006, Bayesian adaptive — (1-Posterior probability of meeting performance goal given the data)

2. Secondary Outcome: False Lumen Thrombosis
Description: Number of participants with partial or complete False Lumen Thrombosis in the region of the aorta covered by the Conformable TAG device.
Time Frame: Last available follow-up through 5 years
Population: Participants with contrast-enhanced CT imagery performed during the specified follow-up period were included in this analysis
Measure: Number; unit: participants
Arm/Group | GORE Conformable TAG® Device Surgical Implant
Number analyzed (Participants) | 45
participants
  Complete Thrombosis | 38
  Partial Thrombosis | 6
  Unknown | 1

3. Secondary Outcome: Aortic Rupture
Description: Number of participants with thoracic aortic rupture
Time Frame: Last available follow-up through 5 years
Measure: Number; unit: participants
Arm/Group | GORE Conformable TAG® Device Surgical Implant
Number analyzed (Participants) | 50
participants | 2

4. Secondary Outcome: Additional Dissection Based Intervention Rate
Description: Number of participants that required additional dissection-based interventions defined as interventions related to malperfusion, rupture, or both, as adjudicated by CEC or Sponsor. Additional dissection based interventions included: peripheral stenting, fenestration, implantation of additional endovascular stent-grafts or other surgeries.
Time Frame: Last available follow-up through 5 years
Measure: Number; unit: participants
Arm/Group | GORE Conformable TAG® Device Surgical Implant
Number analyzed (Participants) | 50
participants | 9

5. Primary Outcome: Exclusion of Primary Entry Tear
Description: Number of subjects with successful coverage of Primary Entry Tear as assessed by the Core Lab using contrast-enhanced CT imagery
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | GORE Conformable TAG® Device Surgical Implant
Number analyzed (Participants) | 40
participants | 39

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | GORE Conformable TAG® Device Surgical Implant
All-Cause Mortality (participants affected / at risk) | 13/50
Serious Adverse Events (participants affected / at risk) | 38/50
Other Adverse Events (participants affected / at risk) | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GORE Conformable TAG® Device Surgical Implant (N=50)
Anaemia (Blood and lymphatic system disorders) | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 6
Atrial fibrillation (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 3
Cardio-respiratory arrest (Cardiac disorders) | 2
Cardiogenic shock (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Complication of device removal (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 4
Stent-graft endoleak (General disorders) | 6
Ischaemic hepatitis (Hepatobiliary disorders) | 1
Abdominal wall abscess (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Groin infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia pseudomonal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Incision site oedema (Injury, poisoning and procedural complications) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Troponin increased (Investigations) | 1
White blood cell count increased (Investigations) | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Alcoholic seizure (Nervous system disorders) | 1
Basal ganglia infarction (Nervous system disorders) | 1
Brain injury (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Carotid artery dissection (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 4
Encephalopathy (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Monoplegia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Spinal cord infarction (Nervous system disorders) | 1
Spinal cord ischaemia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Unresponsive to stimuli (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Delirium tremens (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Anuria (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Renal atrophy (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8
Accelerated hypertension (Vascular disorders) | 1
Aortic aneurysm (Vascular disorders) | 2
Aortic aneurysm rupture (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 5
Aortic dissection rupture (Vascular disorders) | 1
Aortic rupture (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
False lumen dilatation of aortic dissection (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 2
Labile blood pressure (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral artery stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GORE Conformable TAG® Device Surgical Implant (N=50)
Anaemia (Blood and lymphatic system disorders) | 10
Leukocytosis (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Angina pectoris (Cardiac disorders) | 5
Atrial fibrillation (Cardiac disorders) | 6
Bradycardia (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 3
Pericardial effusion (Cardiac disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Oedema peripheral (General disorders) | 8
Peripheral swelling (General disorders) | 3
Pyrexia (General disorders) | 8
Stent-graft endoleak (General disorders) | 6
Cellulitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 8
Device deployment issue (Injury, poisoning and procedural complications) | 3
Blood creatinine increased (Investigations) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypernatraemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 5
Depression (Psychiatric disorders) | 3
Mental status changes (Psychiatric disorders) | 3
Renal failure (Renal and urinary disorders) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 13
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 23
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4
Haematoma (Vascular disorders) | 3
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of less than 90 days. Each investigator will postpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating sites.